CLINICAL TRIAL: NCT01324830
Title: An Open Label Phase Ia/Ib Study of Two Dosing Schedules of BI 847325, Orally Administered Once a Day in Patients With Advanced Solid Tumours, With Repeated Cyclic Administration in Patients With Clinical Benefit
Brief Title: Monotherapy Dose Finding With BI 847325 in Solid Tumours
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1287.1; 2010-023832-18 (EudraCT Number: EudraCT)
Record Dates: First submitted 2011-03-23; First posted 2011-03-29 (Estimated); Results first posted 2018-12-21 (Actual); Last update posted 2018-12-21 (Actual); Status verified 2018-06

CONDITIONS: Neoplasms
MeSH Terms: conditions — Neoplasms

ARMS (2):
- arm A (Experimental): 14 days once a day oral intake of BI 847325 followed by 7 days break in 3-week cycles
  Interventions: Drug: day 1 to day 14
- arm B (Experimental): 5 days once daily oral intake of BI 847325 followed by 2 days break, repeated every week
  Interventions: Drug: day 1 to day 5

INTERVENTIONS:
Drug: day 1 to day 5 — low to high dose
  Arms: arm B
Drug: day 1 to day 14 — low to high dose
  Arms: arm A

SUMMARY:
The aim of the Phase Ia (dose escalation) part of this trial is to assess the maximum tolerated dose (MTD) of BI 847325 administered at escalating doses in 2 treatment arms. In the Phase Ib expansion part of the trial, the aim is to further evaluate the safety profile of BI 847325 at the recommended dose and schedule and to assess target modulation and the potential antitumour efficacy in patients with selected tumour types.

ELIGIBILITY:
Inclusion criteria:

1. Patients with a histologically or cytologically confirmed diagnosis of an advanced unresectable and/or metastatic solid tumour, and who have failed conventional treatment or for whom no therapy of proven efficacy exists or who are not amenable to standard therapies.
2. Age 18 years and older
3. Written informed consent consistent with International conference on harmonization - Good clinical practice (ICH-GCP) and local legislation
4. Eastern Cooperative Oncology Group (ECOG) performance score 0 or 1.
5. Recovery of therapy-related toxicities from previous anti-tumour therapies to Common Terminology Criteria for Adverse Events (CTCAE) = grade 1 (with the exception of alopecia).
6. Written informed consent to the use of archival tumour sample for determination of the BRAF/Tat sarcoma viral oncogene homolog (RAS) mutational status.
7. Life expectancy of at least 12 weeks.
8. In escalation phase, when pharmacokinetic (PK) close to predicted Cmax or when signs of progressive disease (PD) modulation present, optional tumour biopsies (at same timepoints as in expansion phase) for the patients who consented to it.

   In addition, all patients included in the expansion phase (part Ib) must:
9. have been diagnosed with one of the following tumours: melanoma, colorectal carcinoma, Non Small Cell Lung Cancer (NSCLC) or exocrine pancreas adenocarcinoma, and have been shown on their archival tumour sample to have KRAS or BRAF mutation.
10. have a measurable disease.
11. have documented/proven progressive disease within the last 6 months, according to Response Evaluation Criteria In Solid Tumours (RECIST) criteria

11. have a tumour lesion accessible for biopsies (pre- and post-treatment): this is mandatory for patients with colorectal carcinoma or melanoma, optional for patients with NSCLC or exocrine pancreas adenocarcinoma.

Exclusion criteria:

1. Inability to swallow tablets.
2. Additional other serious illness , concomitant non-oncological disease (e.g. active infectious disease or known chronic Hepatitis B/Hepatitis C infection and HIV), or ongoing toxicity from prior therapies considered by the investigator to potentially compromise patient's safety in this trial.
3. Clinical evidence of symptomatic progressive brain or leptomeningeal disease during the last 28 days.
4. Second malignancy currently requiring another anti-cancer therapy.
5. Absolute neutrophil count less than 1500/mm3.
6. Platelet count less than 100 000/mm3.
7. Bilirubin greater than 1.5 mg/dL (>26 µmol/L, Système international (SI) unit equivalent) (except known Gilbert's syndrome).
8. Aspartate amino transferase (AST) and/or alanine amino transferase (ALT) greater than 2.5 times the upper limit of normal (if related to liver metastases, greater than five times the upper limit of normal).
9. Serum creatinine greater than 1.5 mg/dL (>132 µmol/L, SI unit equivalent).
10. Previous episode of QT prolongation due to a medication which, as a result of it, had to be discontinued; or long QT syndrome; or corrected QT interval (QTc) with Fridericia's correction >480 msec on screening ECG.
11. Pregnancy or breastfeeding.
12. Women or men who are sexually active and unwilling to use a medically acceptable method of contraception.
13. Treatment with other investigational drugs or participation in another clinical interventional trial within the past four weeks before start of therapy or concomitant with this trial.
14. Systemic anti-cancer therapy or radiotherapy within the past four weeks before start of therapy or concomitantly with this trial. This restriction does not apply to Luteinizing hormone-releasing hormone (LHRH) agonists, steroids and bisphosphonates.
15. Patients unable to comply with the protocol.
16. Active alcohol or drug abuse.
17. history or presence of cardiovascular abnormalities deemed clinically relevant by the investigator. Myocardial infarction within 6 months prior to study.
18. Cardiac left ventricular ejection fraction <50% or less than institutional lower limit of normal by Multiple Gated Acquisition scan (MUGA) or echocardiography

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2011-04-15 (Actual); Primary Completion 2013-06-06 (Actual); Study Completion 2013-10-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (2):
- Belgium (2):
  - 1287.1.3201 Boehringer Ingelheim Investigational Site, Brussels
  - 1287.1.3202 Boehringer Ingelheim Investigational Site, Leuven

RESULTS

PARTICIPANT FLOW:
Groups:
- Schedule A BI 847325 6 mg (A1): Schedule A BI 847325 6 mg/day group. Schedule A: 2 weeks on treatment, 1 week off treatment, repeated every 3 weeks. BI 847325 tablet(s) administered once daily in the morning 1 hour before breakfast and taken with at least 250 mL of water.
- Schedule A BI 847325 9 mg (A2): Schedule A BI 847325 9 mg/day group. Schedule A: 2 weeks on treatment, 1 week off treatment, repeated every 3 weeks. BI 847325 tablet(s) administered once daily in the morning 1 hour before breakfast and taken with at least 250 mL of water.
- Schedule A BI 847325 13 mg (A3): Schedule A BI 847325 13 mg/day group. Schedule A: 2 weeks on treatment, 1 week off treatment, repeated every 3 weeks. BI 847325 tablet(s) administered once daily in the morning 1 hour before breakfast and taken with at least 250 mL of water.
- Schedule A BI 847325 19 mg (A4): Schedule A BI 847325 19 mg/day group. Schedule A: 2 weeks on treatment, 1 week off treatment, repeated every 3 weeks. BI 847325 tablet(s) administered once daily in the morning 1 hour before breakfast and taken with at least 250 mL of water.
- Schedule A BI 847325 26 mg (A5): Schedule A BI 847325 26 mg/day group. Schedule A: 2 weeks on treatment, 1 week off treatment, repeated every 3 weeks. BI 847325 tablet(s) administered once daily in the morning 1 hour before breakfast and taken with at least 250 mL of water.
- Schedule A BI 847325 33 mg (A6): Schedule A BI 847325 33 mg/day group. Schedule A: 2 weeks on treatment, 1 week off treatment, repeated every 3 weeks. BI 847325 tablet(s) administered once daily in the morning 1 hour before breakfast and taken with at least 250 mL of water.
- Schedule A BI 847325 46 mg (A7): Schedule A BI 847325 46 mg/day group. Schedule A: 2 weeks on treatment, 1 week off treatment, repeated every 3 weeks. BI 847325 tablet(s) administered once daily in the morning 1 hour before breakfast and taken with at least 250 mL of water.
- Schedule A BI 847325 63 mg (A8): Schedule A BI 847325 63 mg/day group. Schedule A: 2 weeks on treatment, 1 week off treatment, repeated every 3 weeks. BI 847325 tablet(s) administered once daily in the morning 1 hour before breakfast and taken with at least 250 mL of water.
- Schedule A BI 847325 86 mg (A9): Schedule A BI 847325 86 mg/day group. Schedule A: 2 weeks on treatment, 1 week off treatment, repeated every 3 weeks. BI 847325 tablet(s) administered once daily in the morning 1 hour before breakfast and taken with at least 250 mL of water.
- Schedule A BI 847325 120 mg (A10): Schedule A BI 847325 120 mg/day group. Schedule A: 2 weeks on treatment, 1 week off treatment, repeated every 3 weeks. BI 847325 tablet(s) administered once daily in the morning 1 hour before breakfast and taken with at least 250 mL of water.
- Schedule A BI 847325 160 mg (A11): Schedule A BI 847325 160 mg/day group. Schedule A: 2 weeks on treatment, 1 week off treatment, repeated every 3 weeks. BI 847325 tablet(s) administered once daily in the morning 1 hour before breakfast and taken with at least 250 mL of water.
- Schedule B BI 847325 6 mg (B1): Schedule B BI 847325 6 mg/day group. Schedule B: 5 days on treatment, 2 days off treatment, repeated every week, in 3-week cycles. BI 847325 tablet(s) administered once daily in the morning 1 hour before breakfast and taken with at least 250 mL of water.
- Schedule B BI 847325 12 mg (B2): Schedule B BI 847325 12 mg/day group. Schedule B: 5 days on treatment, 2 days off treatment, repeated every week, in 3-week cycles. BI 847325 tablet(s) administered once daily in the morning 1 hour before breakfast and taken with at least 250 mL of water.
- Schedule B BI 847325 23 mg (B3): Schedule B BI 847325 23 mg/day group. Schedule B: 5 days on treatment, 2 days off treatment, repeated every week, in 3-week cycles. BI 847325 tablet(s) administered once daily in the morning 1 hour before breakfast and taken with at least 250 mL of water.
- Schedule B BI 847325 46 mg (B4): Schedule B BI 847325 46 mg/day group. Schedule B: 5 days on treatment, 2 days off treatment, repeated every week, in 3-week cycles. BI 847325 tablet(s) administered once daily in the morning 1 hour before breakfast and taken with at least 250 mL of water.
- Schedule B BI 847325 90 mg (B5): Schedule B BI 847325 90 mg/day group. Schedule B: 5 days on treatment, 2 days off treatment, repeated every week, in 3-week cycles. BI 847325 tablet(s) administered once daily in the morning 1 hour before breakfast and taken with at least 250 mL of water.
- Schedule B BI 847325 180 mg (B6): Schedule B BI 847325 180 mg/day group. Schedule B: 5 days on treatment, 2 days off treatment, repeated every week, in 3-week cycles. BI 847325 tablet(s) administered once daily in the morning 1 hour before breakfast and taken with at least 250 mL of water.
- Schedule B BI 847325 130 mg (B7): Schedule B BI 847325 130 mg/day group. Schedule B: 5 days on treatment, 2 days off treatment, repeated every week, in 3-week cycles. BI 847325 tablet(s) administered once daily in the morning 1 hour before breakfast and taken with at least 250 mL of water.
- Schedule B BI 847325 150 mg (B8): Schedule B BI 847325 150 mg/day group. Schedule B: 5 days on treatment, 2 days off treatment, repeated every week, in 3-week cycles. BI 847325 tablet(s) administered once daily in the morning 1 hour before breakfast and taken with at least 250 mL of water.
Period: Overall Study
Arm/Group | Schedule A BI 847325 6 mg (A1) | Schedule A BI 847325 9 mg (A2) | Schedule A BI 847325 13 mg (A3) | Schedule A BI 847325 19 mg (A4) | Schedule A BI 847325 26 mg (A5) | Schedule A BI 847325 33 mg (A6) | Schedule A BI 847325 46 mg (A7) | Schedule A BI 847325 63 mg (A8) | Schedule A BI 847325 86 mg (A9) | Schedule A BI 847325 120 mg (A10) | Schedule A BI 847325 160 mg (A11) | Schedule B BI 847325 6 mg (B1) | Schedule B BI 847325 12 mg (B2) | Schedule B BI 847325 23 mg (B3) | Schedule B BI 847325 46 mg (B4) | Schedule B BI 847325 90 mg (B5) | Schedule B BI 847325 180 mg (B6) | Schedule B BI 847325 130 mg (B7) | Schedule B BI 847325 150 mg (B8)
Started | 3 | 3 | 3 | 3 | 7 | 7 | 3 | 3 | 5 | 6 | 4 | 1 | 1 | 1 | 1 | 3 | 3 | 6 | 6
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 3 | 3 | 3 | 3 | 7 | 7 | 3 | 3 | 5 | 6 | 4 | 1 | 1 | 1 | 1 | 3 | 3 | 6 | 6
Not completed — Progressive Disease | 3 | 2 | 3 | 3 | 6 | 6 | 3 | 3 | 3 | 6 | 2 | 1 | 1 | 1 | 1 | 3 | 2 | 3 | 4
Not completed — Dose limiting toxicity | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1
Not completed — Reason not mentioned above | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Adverse Event, serious fatal | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event, non-fatal | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Treated Set (TS): included all patients who were documented to have received and taken at least one BI 847325 dose.
Groups:
- Total: Total of all reporting groups
Arm/Group | Schedule A BI 847325 6 mg (A1) | Schedule A BI 847325 9 mg (A2) | Schedule A BI 847325 13 mg (A3) | Schedule A BI 847325 19 mg (A4) | Schedule A BI 847325 26 mg (A5) | Schedule A BI 847325 33 mg (A6) | Schedule A BI 847325 46 mg (A7) | Schedule A BI 847325 63 mg (A8) | Schedule A BI 847325 86 mg (A9) | Schedule A BI 847325 120 mg (A10) | Schedule A BI 847325 160 mg (A11) | Schedule B BI 847325 6 mg (B1) | Schedule B BI 847325 12 mg (B2) | Schedule B BI 847325 23 mg (B3) | Schedule B BI 847325 46 mg (B4) | Schedule B BI 847325 90 mg (B5) | Schedule B BI 847325 180 mg (B6) | Schedule B BI 847325 130 mg (B7) | Schedule B BI 847325 150 mg (B8) | Total
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 7 | 7 | 3 | 3 | 5 | 6 | 4 | 1 | 1 | 1 | 1 | 3 | 3 | 6 | 6 | 69
Age, Continuous [Mean (Standard Deviation); unit: Years] | 58.7 (8.1) | 62.7 (3.5) | 58.7 (4.2) | 57.7 (12.2) | 58.9 (9.8) | 55.3 (14.1) | 66 (10.4) | 55.3 (5.1) | 58.6 (9.9) | 59.3 (8.2) | 55 (7.4) | 60 (0) | 49 (0) | 44 (0) | 62 (0) | 49.3 (15.3) | 42.7 (3.5) | 62.2 (13.5) | 51.7 (13.4) | 56.8 (10.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 1 | 1 | 5 | 3 | 2 | 0 | 3 | 1 | 3 | 0 | 1 | 0 | 1 | 1 | 2 | 3 | 4 | 36
  Male | 1 | 0 | 2 | 2 | 2 | 4 | 1 | 3 | 2 | 5 | 1 | 1 | 0 | 1 | 0 | 2 | 1 | 3 | 2 | 33

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients With Dose Limiting Toxicity During the First Treatment Cycle in Phase Ia Part of the Study
Description: Occurrence of dose limiting toxicity (DLT) during the first treatment cycle for the treatment Schedules A and B.
  Some patients excluded from Treated Set (TS) as they were not evaluable for determination of maximum tolerated dose. Thus the number of evaluable TS patients are not the same as the number of original TS patients.
Time Frame: 3 weeks
Population: Treated Set (TS)
Measure: Number; unit: Percentage of participants
Groups:
- Schedule A Total (Total A): All patients with schedule A. Schedule A: 2 weeks on treatment, 1 week off treatment, repeated every 3 weeks.
- Schedule B Total (Total B): Schedule B total treated patients. Schedule B: 5 days on treatment, 2 days off treatment, repeated every week, in 3-week cycles.
- Total Patients: Schedule A and B total patients.
Arm/Group | Schedule A BI 847325 6 mg (A1) | Schedule A BI 847325 9 mg (A2) | Schedule A BI 847325 13 mg (A3) | Schedule A BI 847325 19 mg (A4) | Schedule A BI 847325 26 mg (A5) | Schedule A BI 847325 33 mg (A6) | Schedule A BI 847325 46 mg (A7) | Schedule A BI 847325 63 mg (A8) | Schedule A BI 847325 86 mg (A9) | Schedule A BI 847325 120 mg (A10) | Schedule A BI 847325 160 mg (A11) | Schedule B BI 847325 6 mg (B1) | Schedule B BI 847325 12 mg (B2) | Schedule B BI 847325 23 mg (B3) | Schedule B BI 847325 46 mg (B4) | Schedule B BI 847325 90 mg (B5) | Schedule B BI 847325 180 mg (B6) | Schedule B BI 847325 130 mg (B7) | Schedule B BI 847325 150 mg (B8) | Schedule A Total (Total A) | Schedule B Total (Total B) | Total Patients
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 6 | 6 | 3 | 3 | 3 | 6 | 3 | 1 | 1 | 1 | 1 | 3 | 3 | 6 | 6 | 42 | 22 | 64
Percentage of participants | 0 | 0 | 0 | 0 | 16.7 | 16.7 | 0 | 0 | 0 | 16.7 | 66.7 | 0 | 0 | 0 | 0 | 0 | 66.7 | 16.7 | 16.7 | 11.9 | 18.2 | 14.1

2. Secondary Outcome: Best Overall Response
Description: Best overall response was the best response a patient experienced during their time on study from the start of treatment until: disease progression, the last evaluable assessment in the absence of progression, or the start of subsequent anti-cancer therapy. Death was not considered as progressive disease when determining best overall response; patients who died prior to an evaluable imaging assessment were reported as not evaluable. Some patients were excluded from TS as they were not evaluable for determination of maximum tolerated dose. Thus the number of evaluable TS patients are not the same as the number of original TS patients.
Time Frame: From the start of treatment until the last evaluable assessment. The data cut-off date is 29-Nov-2013
Population: TS
Measure: Number; unit: Participants
Arm/Group | Schedule A BI 847325 6 mg (A1) | Schedule A BI 847325 9 mg (A2) | Schedule A BI 847325 13 mg (A3) | Schedule A BI 847325 19 mg (A4) | Schedule A BI 847325 26 mg (A5) | Schedule A BI 847325 33 mg (A6) | Schedule A BI 847325 46 mg (A7) | Schedule A BI 847325 63 mg (A8) | Schedule A BI 847325 86 mg (A9) | Schedule A BI 847325 120 mg (A10) | Schedule A BI 847325 160 mg (A11) | Schedule B BI 847325 6 mg (B1) | Schedule B BI 847325 12 mg (B2) | Schedule B BI 847325 23 mg (B3) | Schedule B BI 847325 46 mg (B4) | Schedule B BI 847325 90 mg (B5) | Schedule B BI 847325 180 mg (B6) | Schedule B BI 847325 130 mg (B7) | Schedule B BI 847325 150 mg (B8) | Schedule A Total (Total A) | Schedule B Total (Total B) | Total Patients
Number analyzed (Participants) | 3 | 2 | 3 | 3 | 7 | 7 | 3 | 3 | 5 | 6 | 4 | 1 | 1 | 1 | 1 | 3 | 3 | 6 | 6 | 47 | 22 | 69
Participants
  complete response | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  partial response | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
  stable disease | 0 | 0 | 1 | 1 | 3 | 1 | 0 | 1 | 1 | 2 | 1 | 0 | 0 | 0 | 0 | 2 | 2 | 4 | 2 | 11 | 10 | 21
  progressive disease | 3 | 2 | 2 | 2 | 2 | 4 | 3 | 1 | 2 | 3 | 0 | 1 | 1 | 1 | 1 | 1 | 0 | 1 | 4 | 24 | 10 | 34
  not evaluable | 0 | 1 | 0 | 0 | 2 | 2 | 0 | 1 | 2 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 11 | 2 | 13

3. Secondary Outcome: Objective Response
Description: Objective response was a best overall response of complete or partial response, recorded between the start of treatment and the earliest of disease progression, death, or the end of treatment.
  Some patients excluded from TS as they were not evaluable for determination of maximum tolerated dose. Thus the number of evaluable TS patients are not the same as the number of original TS patients.
Time Frame: From the start of treatment and the earliest of disease progression, death, or the end of treatment. The data cut-off date is 29-Nov-2013.
Population: TS
Measure: Number; unit: Participants
Arm/Group | Schedule A BI 847325 6 mg (A1) | Schedule A BI 847325 9 mg (A2) | Schedule A BI 847325 13 mg (A3) | Schedule A BI 847325 19 mg (A4) | Schedule A BI 847325 26 mg (A5) | Schedule A BI 847325 33 mg (A6) | Schedule A BI 847325 46 mg (A7) | Schedule A BI 847325 63 mg (A8) | Schedule A BI 847325 86 mg (A9) | Schedule A BI 847325 120 mg (A10) | Schedule A BI 847325 160 mg (A11) | Schedule B BI 847325 6 mg (B1) | Schedule B BI 847325 12 mg (B2) | Schedule B BI 847325 23 mg (B3) | Schedule B BI 847325 46 mg (B4) | Schedule B BI 847325 90 mg (B5) | Schedule B BI 847325 180 mg (B6) | Schedule B BI 847325 130 mg (B7) | Schedule B BI 847325 150 mg (B8) | Schedule A Total (Total A) | Schedule B Total (Total B) | Total Patients
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 7 | 7 | 3 | 3 | 5 | 6 | 4 | 1 | 1 | 1 | 1 | 1 | 3 | 6 | 6 | 47 | 22 | 69
Participants
  Objective response: No | 3 | 3 | 3 | 3 | 7 | 7 | 3 | 3 | 5 | 6 | 3 | 1 | 1 | 1 | 1 | 3 | 3 | 6 | 6 | 46 | 22 | 68
  Objective response: Yes | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1

4. Secondary Outcome: Disease Control
Description: Disease control was a best overall response of complete response, partial response or stable disease, recorded between the start of treatment and the earliest of disease progression, death, or the end of treatment. Some patients excluded from TS as they were not evaluable for determination of maximum tolerated dose. Thus the number of evaluable TS patients are not the same as the number of original TS patients.
Time Frame: From the start of treatment to the earliest of disease progression, death, or the end of treatment. The data cut-off date is 29-Nov-2013.
Population: TS
Measure: Number; unit: Participants
Arm/Group | Schedule A BI 847325 6 mg (A1) | Schedule A BI 847325 9 mg (A2) | Schedule A BI 847325 13 mg (A3) | Schedule A BI 847325 19 mg (A4) | Schedule A BI 847325 26 mg (A5) | Schedule A BI 847325 33 mg (A6) | Schedule A BI 847325 46 mg (A7) | Schedule A BI 847325 63 mg (A8) | Schedule A BI 847325 86 mg (A9) | Schedule A BI 847325 120 mg (A10) | Schedule A BI 847325 160 mg (A11) | Schedule B BI 847325 6 mg (B1) | Schedule B BI 847325 12 mg (B2) | Schedule B BI 847325 23 mg (B3) | Schedule B BI 847325 46 mg (B4) | Schedule B BI 847325 90 mg (B5) | Schedule B BI 847325 180 mg (B6) | Schedule B BI 847325 130 mg (B7) | Schedule B BI 847325 150 mg (B8) | Schedule A Total (Total A) | Schedule B Total (Total B) | Total Patients
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 7 | 7 | 3 | 3 | 5 | 6 | 4 | 1 | 1 | 1 | 1 | 1 | 3 | 6 | 6 | 47 | 22 | 69
Participants
  Disease control: No | 3 | 3 | 2 | 2 | 4 | 6 | 3 | 2 | 4 | 4 | 2 | 1 | 1 | 1 | 1 | 1 | 1 | 2 | 4 | 35 | 12 | 47
  Disease control: Yes | 0 | 0 | 1 | 1 | 3 | 1 | 0 | 1 | 1 | 2 | 2 | 0 | 0 | 0 | 0 | 2 | 2 | 4 | 2 | 12 | 10 | 22

ADVERSE EVENTS:
Time Frame: From the start date of trial medication up to 21 days after the last administration of BI 847325, up to 266 days
Arm/Group | Schedule A BI 847325 6 mg (A1) | Schedule A BI 847325 9 mg (A2) | Schedule A BI 847325 13 mg (A3) | Schedule A BI 847325 19 mg (A4) | Schedule A BI 847325 26 mg (A5) | Schedule A BI 847325 33 mg (A6) | Schedule A BI 847325 46 mg (A7) | Schedule A BI 847325 63 mg (A8) | Schedule A BI 847325 86 mg (A9) | Schedule A BI 847325 120 mg (A10) | Schedule A BI 847325 160 mg (A11) | Schedule A Total (Total A) | Schedule B BI 847325 6 mg (B1) | Schedule B BI 847325 12 mg (B2) | Schedule B BI 847325 23 mg (B3) | Schedule B BI 847325 46 mg (B4) | Schedule B BI 847325 90 mg (B5) | Schedule B BI 847325 180 mg (B6) | Schedule B BI 847325 130 mg (B7) | Schedule B BI 847325 150 mg (B8) | Schedule B Total (Total B) | Total Patients
Serious Adverse Events (participants affected / at risk) | 1/3 | 1/3 | 0/3 | 1/3 | 5/7 | 3/7 | 1/3 | 0/3 | 4/5 | 2/6 | 4/4 | 22/47 | 1/1 | 0/1 | 0/1 | 0/1 | 1/3 | 2/3 | 4/6 | 1/6 | 9/22 | 31/69
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 3/3 | 2/3 | 7/7 | 7/7 | 3/3 | 3/3 | 5/5 | 6/6 | 4/4 | 46/47 | 1/1 | 1/1 | 1/1 | 1/1 | 3/3 | 3/3 | 6/6 | 6/6 | 22/22 | 68/69
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Schedule A BI 847325 6 mg (A1) (N=3) | Schedule A BI 847325 9 mg (A2) (N=3) | Schedule A BI 847325 13 mg (A3) (N=3) | Schedule A BI 847325 19 mg (A4) (N=3) | Schedule A BI 847325 26 mg (A5) (N=7) | Schedule A BI 847325 33 mg (A6) (N=7) | Schedule A BI 847325 46 mg (A7) (N=3) | Schedule A BI 847325 63 mg (A8) (N=3) | Schedule A BI 847325 86 mg (A9) (N=5) | Schedule A BI 847325 120 mg (A10) (N=6) | Schedule A BI 847325 160 mg (A11) (N=4) | Schedule A Total (Total A) (N=47) | Schedule B BI 847325 6 mg (B1) (N=1) | Schedule B BI 847325 12 mg (B2) (N=1) | Schedule B BI 847325 23 mg (B3) (N=1) | Schedule B BI 847325 46 mg (B4) (N=1) | Schedule B BI 847325 90 mg (B5) (N=3) | Schedule B BI 847325 180 mg (B6) (N=3) | Schedule B BI 847325 130 mg (B7) (N=6) | Schedule B BI 847325 150 mg (B8) (N=6) | Schedule B Total (Total B) (N=22) | Total Patients (N=69)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 3 | 5
Cardiac tamponade (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Ileus (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Euthanasia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
General physical health deterioration (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 2 | 5
Pain (General disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3
Cholangitis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cholecystitis acute (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Portal vein thrombosis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Drug hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 2
Ejection fraction decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Electrocardiogram ST segment elevation (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Troponin I increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 3 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 4
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Pelvic pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 3
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Schedule A BI 847325 6 mg (A1) (N=3) | Schedule A BI 847325 9 mg (A2) (N=3) | Schedule A BI 847325 13 mg (A3) (N=3) | Schedule A BI 847325 19 mg (A4) (N=3) | Schedule A BI 847325 26 mg (A5) (N=7) | Schedule A BI 847325 33 mg (A6) (N=7) | Schedule A BI 847325 46 mg (A7) (N=3) | Schedule A BI 847325 63 mg (A8) (N=3) | Schedule A BI 847325 86 mg (A9) (N=5) | Schedule A BI 847325 120 mg (A10) (N=6) | Schedule A BI 847325 160 mg (A11) (N=4) | Schedule A Total (Total A) (N=47) | Schedule B BI 847325 6 mg (B1) (N=1) | Schedule B BI 847325 12 mg (B2) (N=1) | Schedule B BI 847325 23 mg (B3) (N=1) | Schedule B BI 847325 46 mg (B4) (N=1) | Schedule B BI 847325 90 mg (B5) (N=3) | Schedule B BI 847325 180 mg (B6) (N=3) | Schedule B BI 847325 130 mg (B7) (N=6) | Schedule B BI 847325 150 mg (B8) (N=6) | Schedule B Total (Total B) (N=22) | Total Patients (N=69)
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 1 | 1 | 2 | 3 | 2 | 2 | 1 | 3 | 3 | 19 | 1 | 0 | 0 | 0 | 0 | 2 | 1 | 5 | 9 | 28
Coagulopathy (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 2 | 3
Lymphopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 3 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 2 | 5
Neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 2 | 6 | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 1 | 5 | 11
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 1 | 0 | 4 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 3 | 7
Atrioventricular block first degree (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1
Supraventricular tachycardia (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Adrenal mass (Endocrine disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Endocrine disorder (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Conjunctivitis (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Diplopia (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Ocular discomfort (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Vision blurred (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 1 | 1 | 2 | 0 | 5 | 7
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 2 | 3
Anal fissure (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1
Anorectal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Ascites (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 2
Colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 2
Constipation (Gastrointestinal disorders) | 1 | 1 | 0 | 1 | 2 | 2 | 2 | 0 | 1 | 2 | 0 | 12 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 3 | 15
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 3 | 0 | 2 | 1 | 4 | 2 | 2 | 16 | 0 | 0 | 0 | 0 | 3 | 2 | 6 | 4 | 15 | 31
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 2 | 3
Faecaloma (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1
Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Mouth ulceration (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 2
Nausea (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 3 | 1 | 0 | 1 | 4 | 3 | 2 | 15 | 0 | 1 | 0 | 0 | 1 | 0 | 4 | 1 | 7 | 22
Oesophagitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 2 | 4
Tooth disorder (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 5 | 0 | 0 | 0 | 2 | 3 | 2 | 14 | 0 | 0 | 0 | 0 | 1 | 1 | 5 | 1 | 8 | 22
Asthenia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 4
Chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Fatigue (General disorders) | 2 | 3 | 1 | 2 | 3 | 4 | 1 | 2 | 2 | 4 | 3 | 27 | 0 | 0 | 1 | 0 | 1 | 0 | 5 | 3 | 10 | 37
General physical health deterioration (General disorders) | 1 | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 0 | 0 | 0 | 5 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5
Oedema (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1
Oedema peripheral (General disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 2 | 0 | 0 | 0 | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4
Pain (General disorders) | 0 | 0 | 2 | 0 | 1 | 2 | 0 | 0 | 0 | 2 | 0 | 7 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 3 | 10
Pyrexia (General disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 1 | 1 | 6 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6
Thrombosis in device (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hepatic pain (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypersensitivity (Immune system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cystitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1
Febrile infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Folliculitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1
Herpes zoster (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1
Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1
Nail infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 2 | 2
Oral herpes (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Rhinitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1
Sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1
Tooth abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 1 | 5 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 6
Vulvovaginal candidiasis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Wound infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1
Pelvic fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1
Radiation alopecia (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Rib fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1
Alanine aminotransferase increased (Investigations) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 0 | 6 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 2 | 8
Amylase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Aspartate aminotransferase increased (Investigations) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 5 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 6
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 4
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Blood creatine phosphokinase increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Blood creatinine increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Blood lactate dehydrogenase increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Electrocardiogram QT prolonged (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1
Haematocrit decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1
Lipase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Lymphocyte count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1
Troponin T increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3
Troponin increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Weight decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 4
Decreased appetite (Metabolism and nutrition disorders) | 1 | 3 | 1 | 1 | 2 | 1 | 1 | 0 | 2 | 2 | 1 | 15 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 1 | 5 | 20
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 2
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 1 | 1 | 1 | 6 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 3 | 9
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 2 | 4
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 3
Hypovitaminosis (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 2 | 4
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1
Balance disorder (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Dysgeusia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 2
Headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 2
Paraesthesia (Nervous system disorders) | 0 | 0 | 1 | 0 | 2 | 1 | 0 | 0 | 0 | 1 | 1 | 6 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 5
Confusional state (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Depression (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2
Dysuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Renal failure (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 2 | 1 | 6 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 3 | 9
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 1 | 4 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 3 | 7
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 2
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Petechiae (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1
Hot flush (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypertension (Vascular disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 4
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1
Intermittent claudication (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1
Lymphoedema (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Vascular compression (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

LIMITATIONS AND CAVEATS:
As the trial was terminated without commencing Phase Ib, the endpoints of progression-free survival, time to objective response, duration of objective response and duration of disease control were specified as further endpoints for Phase Ia.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results.

Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.